CLINICAL TRIAL: NCT02357810
Title: A Phase II Study of Pazopanib With Oral Topotecan in Patients With Metastatic and Non-resectable Soft Tissue and Bone Sarcomas
Brief Title: Pazopanib Hydrochloride and Topotecan Hydrochloride in Treating Patients With Metastatic Soft Tissue and Bone Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: GlaxoSmithKline (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 14S03; NCI-2014-02583 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00200112; NU 14S03 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Adult Liposarcoma; Metastatic Liposarcoma; Metastatic Osteosarcoma; Recurrent Adult Soft Tissue Sarcoma; Recurrent Liposarcoma; Recurrent Osteosarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Liposarcoma; Osteosarcoma; Sarcoma | interventions — pazopanib; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pazopanib hydrochloride, topotecan hydrochloride) (Experimental): Patients receive pazopanib hydrochloride PO QD on days 1-28 and topotecan hydrochloride PO on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pazopanib Hydrochloride; Drug: Oral Topotecan Hydrochloride; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient
Drug: Oral Topotecan Hydrochloride — Given PO
  Other Names: Hycamtin Capsules; Oral Hycamtin
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
The purpose of this clinical research study is to learn if pazopanib when given in combination with topotecan can help to control sarcomas. The safety of this drug combination will also be studied. Pazopanib hydrochloride and topotecan hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine progression free rate at week 12 for patients with soft tissue sarcoma (STS) treated with pazopanib (pazopanib hydrochloride) plus oral topotecan (topotecan hydrochloride).

SECONDARY OBJECTIVES:

I. To determine the overall response rate for patients with STS treated with combination pazopanib and topotecan.

II. To determine the clinical benefit rate (complete response [CR] + partial response [PR] + stable disease [SD]) for patients with STS treated with combination pazopanib and topotecan.

III. To determine median progression-free rate (PFR) for patients with STS treated with combination pazopanib and topotecan.

IV. To evaluate overall survival (OS) for patients with STS treated with combination pazopanib and topotecan.

V. To assess safety and tolerability for patients treated with combination pazopanib and topotecan.

VI. To estimate the PFR for patients with osteosarcoma treated with combination pazopanib and topotecan.

VII. To estimate the PFR for patients with liposarcoma treated with combination pazopanib and topotecan.

TERTIARY OBJECTIVES:

I. To estimate the correlation of PFR and OS to levels of soluble vascular endothelial growth factor receptor 2 (sVEGFR2) and phosphatidylinositol-glycan biosynthesis class F (PIGF).

OUTLINE:

Patients receive pazopanib hydrochloride orally (PO) once daily (QD) on days 1-28 and topotecan hydrochloride PO on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity or until discontinuation per patient preference or physician recommendation.

After completion of study treatment, patients are followed up every 6 months for 2 or 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow-up
* Patients must have a histologically confirmed diagnosis of:

  * Metastatic soft tissue sarcomas (non-liposarcoma)
  * Metastatic osteosarcoma
  * Metastatic liposarcoma- high grade, de-differentiated, or myxoid Note: pathology is not required to be reviewed at the treating institution; a copy of the pathology report is sufficient for eligibility purposes
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patients must have measurable disease within 4 weeks prior to registration by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10mm with spiral computed tomography (CT) scan
* Patients must have had a minimum of 1 and a maximum of 4 prior chemotherapy regimens for recurrent/metastatic disease; it will be up to the investigator to determine what constitutes a "regimen" in each case; the last dose of systemic therapy much have been given at least 4 weeks prior to initiation of therapy; patients receiving BCNU or mitomycin C must have received their last dose at least 6 weeks prior to initiation of therapy
* Patients with brain metastasis are eligible for participation only if they have been treated with definitive surgery or radiation (surgery ± radiotherapy, radiosurgery, or gamma knife) and meet both of the following criteria: a) are asymptomatic and b) have no requirement for steroids or enzyme-inducing anticonvulsants in prior 12 week interval
* Absolute neutrophil count (ANC) >= 1.5 X 10^9/L (tested within 7 days prior to Registration)
* Hemoglobin >= 9 g/dL (5.6 mmol/L)

  * Subjects may not have had a transfusion within 7 days of screening assessment
* Platelets >= 100 X 10^9/L

  * Subjects may not have had a transfusion within 7 days of screening assessment
* Prothrombin time (PT) or international normalized ratio (INR) =< 1.2 X upper limit of normal (ULN)

  * Subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation
* Activated partial thromboplastin time (aPTT) =< 1.2 X ULN
* Total bilirubin =< 1.5 X ULN
* Alanine amino transferase (ALT) and aspartate aminotransferase (AST) =< 2.5 X ULN

  * Concomitant elevations in bilirubin and AST/ALT above 1.0 x ULN (upper limit of normal) are not permitted
* Serum creatinine =< 1.5 mg/dL (133 umol/L) or, if > 1.5 mg/dL: calculated creatinine clearance (ClCR) >= 30 mL/min to >= 50 mL/min
* Urine protein to creatinine ratio (UPC) < 1

  * If UPC >= 1, then a 24-hour urine protein must be assessed; subjects must have a 24-hour urine protein value < 1 g to be eligible; use of urine dipstick for renal function assessment is not acceptable
* Females of child-bearing potential (FOCBP) and males must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 30 days following completion of therapy; should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; Note: a FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy
  * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* FOCBP must have a negative pregnancy test within 7 days prior to registration on study

  * Note: female patients who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug
* Are able to swallow and retain oral tablets

Exclusion Criteria:

* Patients with any of the following sarcoma histologic subtypes will not be eligible for participation:

  * Alveolar soft-part sarcoma
  * Chondrosarcoma
  * Dermatofibrosarcoma
  * Ewing sarcoma
  * Gastrointestinal stromal tumor (GIST)
  * Kaposi sarcoma (non-human immunodeficiency virus [HIV] and HIV related disease)
  * Mixed mesodermal tumor/carcinosarcoma
  * Low grade (grade 1) sarcomas
  * Rhabdomyosarcoma (embryonal, alveolar, pleomorphic)
  * Interdigitating dendritic sarcoma
  * Giant cell tumor of the bone
* Patients must not have received prior treatment with pazopanib or topotecan
* Patients must not have an active secondary malignancy
* Prior malignancy, unless they have been disease-free for 3 years, or have a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

  * Active peptic ulcer disease
  * Known intraluminal metastatic lesion/s with risk of bleeding
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

  * Malabsorption syndrome
  * Major resection of the stomach or small bowel
* Corrected QT interval (QTc) > 480 msecs using Bazett's formula
* History of any one or more of the following cardiovascular conditions within the past 12 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft surgery
  * Symptomatic peripheral vascular disease
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of >= 140 mmHg or diastolic blood pressure (DBP) of >= 90mmHg Note: initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry; following antihypertensive medication initiation or adjustment, blood pressure (BP) must be re-assessed three times at approximately 2-minute intervals; at least 24 hours must have elapsed between anti-hypertensive medication initiation or adjustment and BP measurement; these three values should be averaged to obtain the mean diastolic blood pressure and the mean systolic blood pressure; the mean SBP / DBP ratio must be < 140/90 mmHg (or 150/90 mm Hg, if this criterion deemed safe by principal investigator [PI] and the quality assurance monitor [QAM]) in order for a patient to be eligible for the study
* Patients with a history of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism, or untreated deep venous thrombosis (DVT); patients with DVT must have received appropriate therapy for at least 6 months to be considered eligible
* Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major surgery)
* Evidence of active bleeding or bleeding diathesis
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage

  * Large protruding endobronchial lesions in the main or lobar bronchi are excluded; however, endobronchial lesions in the segmented bronchi are allowed
  * Lesions extensively infiltrating the main or lobar bronchi are excluded; however, minor infiltrations in the wall of the bronchi are allowed
* Recent hemoptysis (>= 1/2 teaspoon [2.5 mL]) of red blood within 8 weeks before first dose of study drug
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with patient's safety, provision of informed consent, or compliance to study procedures
* Unable or unwilling to discontinue use of inducers and inhibitors of cytochrome P450 (CYP450) listed for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study; cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) substrates can be administered, but investigators will need to be aware of possible increased or decreased effectiveness of the non-study drug and this should be recorded in concomitant medications; breast cancer resistance protein (BCRP) and p-glycoprotein (PgP) inducers and inhibitors will be also prohibited
* Treatment with any of the following anti-cancer therapies:

  * Radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of therapy
  * Chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of therapy
* Administration of any non-oncologic investigational drug within 30 days or 5 half-lives whichever is longer prior to receiving the first dose of study treatment
* Any ongoing toxicity related to prior anti-cancer therapy that is > grade 1 and/or that is progressing in severity (exceptions include alopecia, fatigue, and hematologic toxicities)
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib or topotecan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2015-03-21 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Agulnik, Principal Investigator — Northwestern University
Locations (8):
- United States (8):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Northwestern University- Lake Forest Hospital, Lake Forest, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual February 25, 2015 and first patient initiated treatment March 20, 2015. The study was designed to enroll up to 105 patients with soft tissue sarcoma (for at least 92 evauable), up to 36 patients with osteosarcoma and 20 patients with liposarcoma for exploratory data. The study closed to further accrual June 10, 2020.
Pre-assignment Details: All patients reported here signed consent, completed eligibility requirements and were registered to the study.
Period: Registered and Started Treatment
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Started | 178
Signed Consent | 178
Registered to Study | 152
Initiated Treatment on Study | 151
Completed | 151
Not Completed | 27
Not completed — Withdrawal by Subject | 1
Not completed — Found not to be eligible for the study | 26
Period: Reached 12 Weeks Response
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Started | 151
Completed 4 Weeks/1 Cycle | 151
Reached 6 Week Response (Patients assessed as having progression at 6 weeks, discontinue study treatment per protocol.) | 129
Reached 12 Weeks/3 Cycles | 95
Completed | 95
Not Completed | 56
Not completed — Adverse Event | 5
Not completed — Progressive Disease | 39
Not completed — Withdrawal by Subject | 8
Not completed — Protocol Violation | 1
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Other | 1
Period: 12 Week Response and Further Treatment
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Started | 95
Assessed for 12 Week Response (Patients assessed as having progression at 12 weeks, discontinue study treatment per protocol.) | 95
Went on to be Treated After Response (Patients continue treatment until progressive disease, toxicity or patient withdrawal.) | 73
Completed | 73
Not Completed | 22
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 1
Not completed — Progressive Disease | 15
Not completed — Wound Complications | 1
Period: Follow-up at Treatment Discontinuation
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Started (Follow-up= 2yrs for patients with progression/5yrs for patients without progression, or until death or reach date 10.12.21) | 151 (All patients that receive at least one dose of study treatment go into follow up phase of the study.)
Completed | 144
Not Completed | 7
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Patients registered to the study are included in baseline patients only. One patient was registered to the study but did not initiate study treatment.
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Number analyzed (Participants) | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 105
  >=65 years | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 144
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 127
  More than one race | 3
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 152
Histology [Number; unit: participants]
  Soft Tissue Sarcoma | 105
  Liposarcoma | 19
  Osteosarcoma | 28

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival at 12 Weeks for Patients With Soft Tissue Sarcoma (STS) Treated With Pazopanib and Oral Topotecan
Description: PFS will be defined from the time of enrollment to the study until progression of disease or death from any cause, as assessed by RECIST 1.1 and measured at 12 weeks after treatment initiation for patients with STS. PFS estimates will be calculated using Kaplan-Meier methods
  Progression is defined as at least a 20% increase in the sum of the Longest Diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Progression must also involve an increase in size of measurable lesions by at least 5 mm, to minimize the possibility that small changes in a small number of target lesions is falsely interpreted as progression.
Time Frame: At 12 weeks from treatment initiation
Population: Only patients with soft tissue sarcoma were eligible for this endpoint. 105 patients enrolled in this trial had soft tissue sarcoma. 1 patient of these 105 was found not to be evaluable.
Measure: Number; unit: percentage of patients progression free
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Number analyzed (Participants) | 104
percentage of patients progression free | 57.5

2. Secondary Outcome: Overall Response Rate (ORR) for Patients With Soft Tissue Sarcoma (STS) Treated With Combination Pazopanib and Topotecan.
Description: ORR is defined as the percentage of patients with Complete Response (CR) plus those with Partial Response (PR) as assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Patients best response to treatment will be used in ORR.
  Complete Response - Disappearance of all target and non target lesions Partial Response - At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD
Time Frame: During treatment, assessed at 6 weeks, 12 weeks, 20 weeks and then every 2 cycles where one cycle = 28 days and range of cycles completed by patients 1-33.
Population: Patients with Soft Tissue Sarcoma treated on study eligible for this endpoint, even if there are major protocol treatment deviations or patients exhibit objective disease progression prior to the end of cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Number analyzed (Participants) | 104
Participants | 7

3. Secondary Outcome: Clinical Benefit Rate (CBR) for Patients With Soft Tissue Sarcoma (STS) Treated With Combination Pazopanib and Topotecan.
Description: CBR is defined as the percentage of patients with Complete Response (CR) plus those with Partial Response (PR) plus those with Stable Disease (SD) as assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Patients best response to treatment will be used in CBR where, in general the following definitions are used:
  Complete Response - Disappearance of all target and non target lesions Partial Response - At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD Stable Disease - Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum LD since the treatment started.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Number analyzed (Participants) | 104
Participants | 66

4. Secondary Outcome: Overall Survival (OS) for Patients With Soft Tissue Sarcoma (STS) Treated With Combination Pazopanib and Topotecan.
Description: OS will be defined from start of study until death from any cause and estimates will be calculated using Kaplan-Meier methods. At time of Kaplan-meier calculations patients included the analysis who have not experienced the event will be censored at the last date of documentation of survival status.
Time Frame: During treatment where one cycle = 28 days and range of cycles completed by patients 1-33, then for 2 years (for patients with progression) and 5 years (for patients without progression) following discontinuation of treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Number analyzed (Participants) | 104
months | 10.94 [9.30 to 18.73]

5. Secondary Outcome: Number of Patients With Significant Adverse Events, Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03
Description: Toxicities will be tabulated and summarized by the number of patients experiencing each toxicity at grade 3 or grade 4
Time Frame: From treatment initiation until 30 days post last treatment, at the beginning of each cycle where 1 cycle=28 days. Range of cycles completed by patients 1-33 cycles
Measure: Number; unit: patients
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Number analyzed (Participants) | 151
patients
  Anemia | 32
  Platelet count decreased | 61
  Decreased neutrophil count | 80
  Hypertension | 35
  Fatigue | 13
  Nausea | 5
  Hyperglycemia | 6
  Diarrhea | 13
  Vomiting | 11
  Anorexia | 3
  Alkaline phosphatase increase | 6
  Hyponatremia | 17
  Hypocalcemia | 1
  Aspartate aminotransferase increased | 6
  Prolonged PTT | 3
  GGT increase | 7
  Abdominal pain | 7
  Hypokalemia | 6
  Dyspnea | 7
  QTc prolongation | 1
  INR increased | 2
  Alanine aminotransferase increase | 8
  Blood bilirubin increased | 2
  Epistaxis | 2
  Creatinine increase | 2
  Mucositis | 1
  Proteinuria | 6

6. Secondary Outcome: Median Progression Free Survival (PFS) for Patients With Soft Tissue Sarcoma (STS) Treated With Combination Pazopanib and Topotecan.
Description: PFS will be defined from the time of enrollment to the study until progression of disease or death from any cause, as assessed by RECIST 1.1. PFS estimates will be calculated using Kaplan-Meier methods. Patients included in the analysis, who did not experiences the event at the time of the calculation were censored from the last documentation of being progression free.
  Progression is defined as at least a 20% increase in the sum of the Longest Diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Progression must also involve an increase in size of measurable lesions by at least 5 mm, to minimize the possibility that small changes in a small number of target lesions is falsely interpreted as progression.
Time Frame: During treatment, assessed at 6 weeks, 12 weeks, 20 weeks and then every 2 cycles where one cycle = 28 days and range of cycles completed by patients 1-33. And then for up to 5 years post treatment discontinuation.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Number analyzed (Participants) | 104
months | 4.37 [3.09 to 6.21]

7. Secondary Outcome: Progression Free Survival in Patients With Osteosarcoma Treated With Combination Pazopanib and Topotecan.
Description: as for outcome 6
Time Frame: During treatment, assessed at 6 weeks, 12 weeks, 20 weeks and then every 2 cycles where one cycle = 28 days and range of cycles completed by patients 1-33. Then for up to 5 years post treatment discontinuation
Population: Only patients with Osteosarcoma were eligible for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Number analyzed (Participants) | 28
months | 4.47 [2.76 to 8.28]

8. Secondary Outcome: Progression Free Survival for Patients With Liposarcoma Treated With Combination Pazopanib and Topotecan.
Description: PFS will be defined from the time of enrollment to the study until progression of disease or death from any cause, as assessed by RECIST 1.1. PFS estimates will be calculated using Kaplan-Meier methods. Patients who did not experiences the event at the time of the calculation were censored from the last documentation of being progression free.
  Progression is defined as at least a 20% increase in the sum of the Longest Diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Progression must also involve an increase in size of measurable lesions by at least 5 mm, to minimize the possibility that small changes in a small number of target lesions is falsely interpreted as progression.
Time Frame: During treatment, assessed at 6 weeks, 12 weeks, 20 weeks and then every 2 cycles where one cycle = 28 days and range of cycles completed by patients 1-33. Then up to 5 years post treatment discontinuation.
Population: Patients with liposarcoma were eligible for this endpoint.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Number analyzed (Participants) | 19
Months | 1.48 [1.25 to 12.85]

9. Other Pre Specified Outcome: Change in Cytokine Levels
Description: Verification of results of Sleijfer et al and to determine if there is an even earlier correlation that can be detected between levels of these cytokines and PFR as well as OS which may allow us to better predict treatment response early on in therapy.
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

10. Post Hoc Outcome: Overall Survival of Patients With Liposarcoma Treated With With Pazopanib and Oral Topotecan Combination
Description: OS is defined from enrollment to the study until death from any cause. OS estimates will be calculated using Kaplan-Meier methods. Patients included in the analysis who did not experience the event at the time of the calculation, were censored from the last documentation of being progression free.
Time Frame: During treatment, where one cycle = 28 days and range of cycles completed by patients 1-33. Then for up to 5 years post treatment discontinuation.
Population: At the time of the calculation, 12 events were seen out of a possible 16.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Number analyzed (Participants) | 16
Weeks | 55.86 [14.57 to 125.00]

11. Post Hoc Outcome: Duration of Best Response in Patients With Soft Tissue Sarcoma Treated With Pazopanib and Topotecan Combination
Description: Duration of response is measured from the time of best response (Complete Response (CR), Partial Response (PR), Stable Disease SD)) as assessed by RECIST v1.1 until time of Progressive Disease (PD). Patients whose best response was PD are removed from this analysis. Patients who are included in the analysis but do not experience the event at the time of the calculation, will be censored at the last known date documented.
  CR-Disappearance of all target and non target lesions PR-≥30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD SD-Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started PD- ≥20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: From time of initial response until progressive disease, up to 60 weeks.
Population: At time of analysis 66 events were seen out of the possible 68.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Number analyzed (Participants) | 68
Weeks | 25.71 [20.00 to 33.29]

12. Post Hoc Outcome: Duration of Best Response in Patients With Liposarcoma Treated With Pazopanib and Topotecan Combination
Description: as for outcome 11
Time Frame: From time of initial response until progressive disease, up to 60 weeks.
Population: At the time of the analysis 7 events were seen out of a possible 8.
Measure: Median (97.5% Confidence Interval); unit: Weeks
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
Number analyzed (Participants) | 8
Weeks | 33.79 [19.14 to 96.86]

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) data was collected for each patient from treatment initiation until 30 days post last treatment, at the beginning of each cycle where 1 cycle=28 days. Range of cycles completed by patients 1-33 cycles. Serious Adverse Event (SAE) data is collected from the time of consent (regardless of if a patient initiates treatment) until 30 days post last treatment. All cause mortality was collected for patients who initiated treatment, and up to 5 years post treatment discontinuation.
Description: Data entry is currently being completed for the most recent patients - this Section will be updated with final adverse event data at the end of the study. Due to data collection methods some SAE data may also be included in Other AE as well as in Serious Adverse Event Section. Patients who signed consent/did not initiate treatment are included as at risk for SAE but not at risk for other AEs due to 5 out of 26 screenfail patients experiencing an SAE.
Arm/Group | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 116/151
Serious Adverse Events (participants affected / at risk) | 88/178
Other Adverse Events (participants affected / at risk) | 151/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride) (N=178)
Renal Calculi (Renal and urinary disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Generalized muscle weakness and malaise (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Upper respiratory infection (Infections and infestations) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Wound complications (Injury, poisoning and procedural complications) | 1 (1)
Urinary track infection with fever (Infections and infestations) | 1 (1)
Increased alkaline phosphatase (Investigations) | 1 (1)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Patient also with bowel obstruction at the time of the event
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Patient also with back pain at the time of the event
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Patient also with Pneumothroax at the time of the event
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Superior Vena Cava Syndrome (Vascular disorders) | 1 (1) — Patient also with neutropenia and fever at the time of the event
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Skin Infection (Infections and infestations) | 2 (2)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient also with dyspnea at the time of the event
Hypotension (Vascular disorders) | 1 (1) — Patient also with pain at the time of the event
Thrombocytopenia (Investigations) | 1 (1)
lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Stroke (Vascular disorders) | 1 (1) — Patient also with Left Ventricular Systolic Dysfunction at the time of the event
Blurred Vision (Eye disorders) | 1 (1) — Patient also with headache at the time of the event
Syncope (Nervous system disorders) | 1 (1) — Patient also with dehydration at the time of the event
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
obstructed biliary stent (Gastrointestinal disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 2 (2) — One patient was a screenfail and did not initiate treatment due to the event
Anemia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Thrombocytopenia (Investigations) | 1 (1) — Patient also with urinary tract obstruction at the time of the event
Nausea and diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea and pain (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
INR increase (Investigations) | 1 (1)
Colonic and bladder perforation (Gastrointestinal disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient was screenfail due to the event and did not initiated treatment
Pain in extremity with anemia (General disorders) | 1 (1) — Patient was screenfail due to the event and did not initiated treatment
Back pain (General disorders) | 2 (2)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypoxemia with dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Abdominal pain and distension (Gastrointestinal disorders) | 1 (1)
Pelvic pain (General disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Respiratory failure with dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea/vomiting/diarrhea (Gastrointestinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (4)
Platelet Count Decrease (Investigations) | 1 (1) — Patietn also with neutrophil count decrease at the time of the event
Dehydration (Gastrointestinal disorders) | 1 (1)
Sepsis with colonic perforation (Gastrointestinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient also with atrial fibrillation at the time of the event
Hematuria (Renal and urinary disorders) | 1 (2)
Edema in limbs (General disorders) | 1 (1) — Patient also with abdominal pain at the time of the event
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — Patient also with diarrhea at the time of the event
Abcess infection (Infections and infestations) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) — Patient also with anemia at the time of the event
Urinary Track infection (Renal and urinary disorders) | 1 (1) — Patient also with back pain and dysuria at the time of the event
Diarrhea (Gastrointestinal disorders) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1) — Patient also with anemia at the time of the event
Back and abdominal pain (General disorders) | 1 (1) — Patient was screenfail due to the event and did not initiated treatment
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient also with fever at the time of the event. Patient was screenfail due to the event and did not initiated treatment
Pancytopenia (Investigations) | 1 (1) — Patient also with neutrophil count decrease and dehydration during this event
Abdominal Abscess/Enterocutaneous Fistula (Gastrointestinal disorders) | 1 (1) — Patient also with febrile neutropenia bilirubin increase and hyponatremia at the time of the event
Elevated liver enzymes and bilirubin (Alkaline phosphatase, ALT, AST, GGT) (Investigations) | 1 (1)
Abdominal abscess and colitis (Gastrointestinal disorders) | 1 (1) — Patient also with sepsis and colvaginal fistula at the time of the event
Pancytopenia (Investigations) | 1 (1) — Patient also with hyponatemia and diarrhea at the time of the event
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Patient also with thromboembolic event and pleural effusion at the time of the event
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pazopanib Hydrochloride, Topotecan Hydrochloride) (N=151)
Anemia (Blood and lymphatic system disorders) | 112
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Leukocytosis (Blood and lymphatic system disorders) | 1
Aortic valve disease (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 6
Heart failure (Cardiac disorders) | 2
Left ventricular systolic dysfunction (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 16
Sinus tachycardia (Cardiac disorders) | 20
Disease progression (Ear and labyrinth disorders) | 4
Ear pain (Ear and labyrinth disorders) | 5
Hearing impaired (Ear and labyrinth disorders) | 1
Middle ear inflammation (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Hyperthyroidism (Endocrine disorders) | 8
Hypothyroidism (Endocrine disorders) | 23
Blurred vision (Eye disorders) | 5
Dry eye (Eye disorders) | 2
Platelet Count Decrease (Eye disorders) | 7
Flashing lights (Eye disorders) | 1
Floaters (Eye disorders) | 5
Photophobia (Eye disorders) | 1
Syncope (Eye disorders) | 1
Watering eyes (Eye disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 44
Bloating (Gastrointestinal disorders) | 4
Colonic fistula (Gastrointestinal disorders) | 1
Colonic hemorrhage (Gastrointestinal disorders) | 1
Heart Failure (Gastrointestinal disorders) | 2
Colonic perforation (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 29
Dental caries (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 87
Dry mouth (Gastrointestinal disorders) | 4
Duodenal ulcer (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 13
Dysphagia (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 9
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 14
Gastrointestinal pain (Gastrointestinal disorders) | 2
Gastroparesis (Gastrointestinal disorders) | 2
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 106
Oral dysesthesia (Gastrointestinal disorders) | 3
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 11
Pancreatitis (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 85
Chills (General disorders) | 3
Death NOS (General disorders) | 3
Edema face (General disorders) | 2
Edema limbs (General disorders) | 22
Edema trunk (General disorders) | 1
Skin Infection (General disorders) | 2
Fatigue (General disorders) | 97
Fever (General disorders) | 18
Flu like symptoms (General disorders) | 6
General disorders and administration site conditions - Other, specify (General disorders) | 26
Irritability (General disorders) | 1
Localized edema (General disorders) | 1
Malaise (General disorders) | 7
Non-cardiac chest pain (General disorders) | 3
Pain (General disorders) | 32
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 1
Anorectal infection (Infections and infestations) | 1
Bronchial infection (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 4
Lip infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 3
Papulopustular rash (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 5
Upper respiratory infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 15
Bruising (Injury, poisoning and procedural complications) | 5
Fall (Injury, poisoning and procedural complications) | 3
Fracture (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Intraoperative endocrine injury (Injury, poisoning and procedural complications) | 1
Urostomy obstruction (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 2
Activated partial thromboplastin time prolonged (Investigations) | 44
Alanine aminotransferase increased (Investigations) | 32
Alkaline phosphatase increased (Investigations) | 48
Aspartate aminotransferase increased (Investigations) | 56
Blood bilirubin increased (Investigations) | 35
Cardiac troponin I increased (Investigations) | 2
Creatinine increased (Investigations) | 16
Ejection fraction decreased (Investigations) | 3
Electrocardiogram QT corrected interval prolonged (Investigations) | 23
GGT increased (Investigations) | 34
INR increased (Investigations) | 26
Investigations - Other, specify (Investigations) | 7
Lymphocyte count decreased (Investigations) | 86
Lymphocyte count increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 116
Pancreatic enzymes decreased (Investigations) | 1
Platelet count decreased (Investigations) | 130
Weight gain (Investigations) | 1
Weight loss (Investigations) | 28
White blood cell decreased (Investigations) | 124
Anorexia (Metabolism and nutrition disorders) | 70
Dehydration (Metabolism and nutrition disorders) | 14
Hypercalcemia (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 78
Hyperkalemia (Metabolism and nutrition disorders) | 8
Hypermagnesemia (Metabolism and nutrition disorders) | 5
Hypernatremia (Metabolism and nutrition disorders) | 3
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 78
Hypocalcemia (Metabolism and nutrition disorders) | 64
Hypoglycemia (Metabolism and nutrition disorders) | 11
Hypokalemia (Metabolism and nutrition disorders) | 46
Hypomagnesemia (Metabolism and nutrition disorders) | 41
Hyponatremia (Metabolism and nutrition disorders) | 56
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 29
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Chest wall pain (Musculoskeletal and connective tissue disorders) | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 20
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18
Trismus (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Dizziness (Nervous system disorders) | 21
Dysarthria (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 31
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 43
Lethargy (Nervous system disorders) | 2
Nervous system disorders - Other, specify (Nervous system disorders) | 4
Neuralgia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 6
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4
Sinus pain (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 6
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 6
Confusion (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 15
Bladder perforation (Renal and urinary disorders) | 1
Bladder spasm (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 15
Proteinuria (Renal and urinary disorders) | 14
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 10
Renal calculi (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 3
Urinary tract obstruction (Renal and urinary disorders) | 3
Urinary tract pain (Renal and urinary disorders) | 3
Urinary urgency (Renal and urinary disorders) | 3
Pelvic pain (Reproductive system and breast disorders) | 3
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 2
Vaginal pain (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 26
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 39
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 6
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 8
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 12
Dry skin (Skin and subcutaneous tissue disorders) | 6
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 16
Pruritus (Skin and subcutaneous tissue disorders) | 4
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 14
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 7
Skin ulceration (Skin and subcutaneous tissue disorders) | 3
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 3
Flushing (Vascular disorders) | 2
Hot flashes (Vascular disorders) | 3
Hypertension (Vascular disorders) | 95
Hypotension (Vascular disorders) | 8
Lymphedema (Vascular disorders) | 3
Superficial thrombophlebitis (Vascular disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT02357810/Prot_SAP_001.pdf